CLINICAL TRIAL: NCT01738074
Title: Phase Three Clinical Trials of Trivalent Rotavirus Genetic Reassortment Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center for Disease Control and Prevention, Henan Province (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: HNCDC-001
Record Dates: First submitted 2012-11-20; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Randomized; Double-blind; Placebo Control Design
Keywords: rotavirus; trivalent genetic reassortment vaccine; Phase three clinical trials

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- trivalent rotavirus genetic reassortment vaccine (Experimental): 2ml of rotavirus genetic reassortment vaccine by mouth every month for three month
  Interventions: Biological: trivalent rotavirus genetic reassortment vaccine
- Placebo (Placebo Comparator): 2ml of placebo by mouth every month for three month
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: trivalent rotavirus genetic reassortment vaccine
  Arms: trivalent rotavirus genetic reassortment vaccine
Biological: Placebo
  Arms: Placebo

SUMMARY:
Assessment and evaluation the rotavirus gastroenteritis prevention effect and severe rotavirus diarrhea reducing effectiveness of human body, which inoculate trivalent rotavirus genetic reassortment vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 13 weeks aged healthy baby;
* Guardian volunteer to participate in the study and sign informed consent;
* have use thermometer as required and the ability to fill in the diary table;
* Subjects guardian can abide by the requirements of clinical research scheme;
* The past has not been vaccinated rotavirus vaccine;
* Normal term eutocia, birth weight up to standard;
* Axillary temperature is 37.0 ℃ or less.

Exclusion Criteria:

* With allergy, convulsion, epilepsy, encephalopathy and spirit history or the family history;
* Be allergy to any ingredients in the vaccine;
* Known immunology function damage or low person;
* Immunosuppressant therapy Accepter;
* Suffering from congenital malformation and developmental disorder;
* Known or suspected also suffer from diseases including: digestive system disease, respiratory system disease, acute infection, mother or I have HIV infection, cardiovascular diseases, malignant tumor during treatment, skin disease;
* Inoculation other vaccine within 7 days.

Ages: 6 Weeks to 13 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10020 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Antibody titer differences in serum | 4 weeks after full vaccination
Incidence differences of rotavirus diarrhea | 2 years after full vaccination.